CLINICAL TRIAL: NCT04156659
Title: A Phase II, Single Arm, Multi-center Trial to Evaluate the Efficacy and Safety of Tisagenlecleucel in Chinese Pediatric and Young Adult Patients With Relapsed or Refractory B-cell Acute Lymphoblastic Leukemia
Brief Title: Study of Tisagenlecleucel in Chinese Pediatric and Young Adult Subjects With Relapsed or Refractory B-cell ALL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was cancelled before enrolling any patients for business related reasons.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTL019B2210
Record Dates: First submitted 2019-10-23; First posted 2019-11-07 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia; ALL; Tisagenlecleucel; CTL019; China
MeSH Terms: conditions — Burkitt Lymphoma | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tisagenlecleucel (Experimental): All patients eligible for treatment with tisagenlecleucel will receive a single dose of tisagenlecleucel.
  For subjects ≤ 50 kg, tisagenlecleucel will be administered as a single infusion of 0.2 to 5.0 x 10^6 CAR positive viable T cells per kg body weight.
  For subjects > 50 kg, tisagenlecleucel will be administered as a single infusion of 0.1 to 2.5 x 10^8 CAR positive viable T cells.
  Interventions: Biological: Tisagenlecleucel

INTERVENTIONS:
Biological: Tisagenlecleucel — A single intravenous (i.v.) infusion of CAR-positive viable T cells.
  Other Names: CTL019

SUMMARY:
This is a single arm, multi-center, phase II study to evaluate the efficacy and safety of tisagenlecleucel in Chinese pediatric and young adult subjects with relapsed or refractory B-cell acute lymphoblastic leukemia (ALL)

DETAILED DESCRIPTION:
The study will have the following sequential phases for all subjects:

* Screening
* Pre-Treatment (Cell Product Preparation and Lymphodepleting Chemotherapy)
* Treatment and Follow-up Tisagenlecleucel infusion should occur within 16 weeks of informed consent. The total duration of the study is 5 years. After tisagenlecluecel infusion, efficacy will be assessed monthly for the first 6 months, then quarterly up to 2 years and semi-annually afterwards up to 5 years, or until the subject relapses.

ELIGIBILITY:
Key Inclusion Criteria:

1. Chinese patients age ≤25 years at the time of informed consent form (ICF) signature.
2. Relapsed or refractory B-cell ALL

   1. 2nd or greater bone marrow (BM) relapse OR
   2. Any BM relapse after allogeneic SCT and must be ≥ 3 months from SCT at the time of screening OR
   3. Primary refractory as defined as not achieving a CR after 2 cycles of a standard first line chemotherapy regimen or chemorefractory as defined by not achieving a CR after 1 cycle of standard chemotherapy for relapsed leukemia OR
   4. Subjects with Ph+ ALL are eligible if they are intolerant to or relapsed/refractory after two lines of tyrosine kinase inhibitor (TKI) therapy, or if TKI therapy is contraindicated OR
   5. Ineligible for allogeneic SCT because of: comorbid disease; other contraindications to allogeneic SCT conditioning regimen; lack of suitable donor; prior SCT; subject declines allogeneic SCT as a therapeutic option after documented discussion about the role of SCT with a BMT physician not part of the study team
3. For relapsed patients, CD19 tumor expression demonstrated in bone marrow or peripheral blood by flow cytometry within 3 months of screening
4. Bone marrow with ≥ 5% lymphoblasts on local morphologic assessment at screening
5. Adequate performance status, cardiac, hepatic, renal and pulmonary function at screening
6. Must meet the institutional criteria to undergo leukapheresis
7. Once all other eligibility criteria are confirmed, must have a leukapheresis material of non-mobilized cells received and accepted for manufacturing.

Key Exclusion Criteria:

1. Isolated extra-medullary disease relapse
2. Subjects with concomitant genetic syndromes associated with bone marrow failure states: such as subjects with Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome. Subjects with Down syndrome will not be excluded.
3. Subjects with Burkitt's lymphoma/leukemia (i.e. subjects with mature B-cell ALL, leukemia with B-cell [sIg positive and kappa or lambda restricted positivity] ALL, with FAB L3 morphology and /or a MYC translocation)
4. Prior anti-CD19 directed therapy, gene therapy or adoptive T cell therapy
5. CNS involvement by ALL, defined as CNS-2 and CNS-3 disease per National Comprehensive Cancer Network guidelines NCCN 2018 v1
6. Active neurological autoimmune or inflammatory disorders (e.g. Guillain-Barre syndrome)
7. History or presence of clinically relevant CNS pathology, e.g., epilepsy, paresis, aphasia, stroke, severe brain injuries, cerebellar disease, organic brain syndrome, or psychosis.
8. Investigational medicinal product within the last 30 days or five half-lives (whichever is longer) prior to screening NOTE: Investigational therapies must not be used at any time while on study until the first progression following tisagenlecleucel infusion.
9. Previous or concurrent malignancy except for curatively treated non-melanoma skin cancers, in situ carcinoma (e.g. cervix, skin), and cancers in complete remission for at least 3 years and without evidence of recurrence

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall Remission Rate (ORR) | From first dosing (single administration, Day 1) up to Month 3
  Evaluate the efficacy of tisagenlecleucel using overall remission rate (ORR) during the 3 months after tisagenlecleucel administration as assessed by the investigator. The ORR is defined as the proportion of subjects with a best overall disease response of Complete Remission (CR) or Complete Remission with Incomplete blood count recovery (CRi)

SECONDARY OUTCOMES:
CR or CRi rate at month 6 | Month 6
  Evaluate the percentage of participants who achieve CR or CRi at Month 6 without SCT after tisagenlecleucel infusion
CR or CRi rate at Day 28 | Day 28
  Evaluate the percentage of participants who achieve CR or CRi at Day 28 after tisagenlecleucel infusion
Best Overall Response (BOR) of CR or CRi with a MRD negative bone marrow | From first dosing (single administration, Day 1) up to Month 3
  Evaluate the percentage of participants who achieve a BOR of CR or CRi with a MRD negative bone marrow during the 3 months after tisagenlecleucel infusion
Duration of remission (DOR) | Average of 60 Months
  DOR, i.e. the time from achievement of CR or CRi, whichever occurs first, to relapse or death due to ALL
Relapse free survival (RFS) | Avarage of 60 Months
  RFS, i.e. the time from achievement of CR or CRi whichever occurs first to relapse or death due to any cause during CR or CRi
Event free survival (EFS) | Average of 60 Months
  EFS, i.e. the time from date of Tisagenlecleucel infusion to the earliest of death, relapse or treatment failure
Overall survival (OS) | Average of 60 Months
  OS, i.e. the time from date of tisagenlecleucel infusion to the date of death due to any reason
Number of Participants with On-Treatments Adverse Events, Serious Adverse Events, and Deaths | From Screening up to Month 60
  Analysis of absolute and relative frequencies for treatment emergent Adverse Event (AE), Serious Adverse Event (SAE) and Deaths by primary System Organ Class (SOC) parameters.
In vivo cellular PK profile of tisagenlecleucel | Up to Month 60
  qPCR and flow cytometry will be used to measure tisagenlecleucel transgene concentration in blood, bone marrow and other matrices/tissues
Serum cytokine | Up to Month 60
  Concentrations of soluble factors (such as IL-10, iFN-y, IL-6) in blood will be summarized by participant and time point
Levels of pre-existing and treatment induced humoral immunogenicity | Up to Month 60
  The humoral immunogenicity assay measures the antibody titers specific to tisagenlecleucel prior to and following infusion
Tociluzumab PK | Up to Day 7 after tocilizumab infusion
  Concentrations of tocilizumab
Levels of prexisting and treatment induced cellular immunogenicity | Up to Month 60
  The cellular immunogenicity assay will assess the presence of T lymphocyte activated by the tisagenlecleucel protein

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com